CLINICAL TRIAL: NCT05500001
Title: Supporting Patients by Family Education in Psychotic Illness: A Prospective Cohort Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other); Families Supporting Adults with Mental Illness-Alberta (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110691
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Psychotic Disorders; Family Members; Anosognosia; Paranoia
Keywords: Young Adult; Psychosis; Family Psychoeducation; Family Burden; Acceptance and Commitment Therapy; LEAP
MeSH Terms: conditions — Psychotic Disorders; Agnosia; Paranoid Disorders

STUDY DESIGN:
Intervention Model Description: A longitudinal pre-post study design will be used. A non-equivalent comparison group will be available for some measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Psychoeducation Intervention Arm (Experimental): These participants will receive the psychoeducation intervention and outcome measures will be taken from them and their young adult service user. The intervention includes psychoeducation on stages of a family's journey, the biopsychosocial basis of psychosis, and skills for coping (Acceptance and Commitment Therapy for Caregivers) and communicating (LEAP).
  Interventions: Behavioral: Supporting Patients by Family Education in Psychotic Illness Group

INTERVENTIONS:
Behavioral: Supporting Patients by Family Education in Psychotic Illness Group — Psychoeducation for families supporting young adults with psychosis.

SUMMARY:
Background: A lack of education, resources, and support for family carers of young adults with psychotic illnesses leaves them ill-equipped to support their loved one. Although family support groups exist, few groups offer evidence-based, skills-focused, psychoeducation taught by certified professionals and provided on a public-health level. By equipping families with skills and knowledge, public healthcare harnesses a powerful ally to maintain community stabilization.

Aims: The primary study goal is to implement a psychoeducation intervention for family carers supporting young adults with psychosis to reduce family burden and foster community stabilization of service users.

Methods: A longitudinal pre-post design will be used to assess the long-term effectiveness of the psychoeducation intervention for family carers supporting a young adult with psychosis on service utilization and functional indexes. Nine expert-reviewed, and family peer-informed psychoeducation modules are administered in 2-hour sessions over 9 weeks to family carers.

Conclusion: Presenting the novel approach of an expert-reviewed, peer-informed psychoeducation intervention for family carers, with a focus on knowledge and skill development, the researchers contribute to literature and best practice in patient and family-centered care.

DETAILED DESCRIPTION:
Background:

A lack of education, resources, and support for family carers of young adults with psychotic illnesses leaves them ill-equipped to support their loved one. Often family carers are excluded from the discharge planning process or are unaware of how to support of their loved one in community. Although best practice documents champion family involvement the implementation of these guidelines is challenge and families are often excluded from care.There is evidence of the disparity between best practice documents and true practice in the literature.

Family inclusion also addresses the impact of psychotic disease on the family's functioning and mental health. Psychotic illness (e.g., anosognosia, paranoia) can interfere with relational health and the natural maturation of family relationships over time. Families face extreme challenges when supporting a young adult with psychotic illness including social isolation, likely because their typical social supports are unable to relate to their situation, prompting them to seek support with those who share their situation (i.e., family support groups). Family carers, even in the face of these hardships, work with great tenacity toward improving service user stability in community.

There is a lack of high-quality effectiveness research showing longitudinal evidence for treatment effects on the carer and the young person in family psychoeducation groups. For example, one study provided a family intervention that was primarily knowledge- and support-based. These researchers used a pre-post design to assess the mental health knowledge, but did not assess long-term effectiveness of the group, overall family functioning, and functioning of the service user.

The intent for this longitudinal pre-post study is to evaluate the effect of skills-based educational programming for family carers supporting young adults admitted to or discharged from hospital with psychosis of any etiology on 6-month and 24-month service user readmission rates and service user/family functional indexes. The investigators hypothesize that system integration of a program which delivers early support for the family carers by way of an educational intervention beginning prior to or shortly after hospital discharge may reduce family burden as well as improve short- and long-term patient outcomes. To the investigators' knowledge, this study is the first to evaluate effectiveness of a family carer skills-based education intervention within a public healthcare system.

The investigators will use a longitudinal pretest-posttest design with a non-equivalent control group to evaluate the short- and long-term effectiveness of this family psychoeducation intervention. While a control group can be used for comparison of the service utilization data for young adults with psychosis using archival data from health records, gathering long-term control group data from families not participating in the trial is unethical in that denial of an intervention for up to two years is potentially harmful to both the families and the young adult they support. Likewise, control group data gathered directly from young adult service users presents the same ethical problem. Using archival health utilization data, however, allows us to exclude any service users' whose families have elected to access the psychoeducation program within the 2-year timeframe of the study. This allows us to find control data for health service utilization while not withholding the psychoeducation intervention from those who seek it. The investigators acknowledge that the control group is non-equivalent because families and service users who chose not to engage in the study may vary systematically from those who did.

Each measure will be taken pre-intervention (i.e., baseline), post-intervention, then again at 6- and 24-months post-intervention. A gift card incentive ($25.00 per data collection meeting) will be provided to family and young adult participants as a token of appreciation for their participation.

Service utilization data will be collected for 12-months pre-intervention to be compared to 12-months post-intervention and 12-24 months post-intervention.

Recruitment:

Study information will be disseminated by clinical teams and through community organizations, and family carers meeting eligibility criteria will self-identify for participation. Once recruited, and with family consent, young adult service users of participating family carers will be contacted for recruitment into the study.

Measures:

A variety of measures will be used to collect functional index data for the family members and the young adult service users. Health utilization data will be mined for 12-months pre-intervention, and up to 24-months post-intervention to assess long term service user outcomes. See Outcome Measures section for details.

Secondary Data Control Group:

While randomization into treatment and control groups was not feasible for this study, non-equivalent control group data can be mined from health records for young adults whose family did not participate in the study.

Intervention:

The educational modules are developed by experts in the areas of interest and are evidence based, family peer-informed and expert peer-reviewed. The curriculum consists of 9 modules delivered weekly over 9 weeks. Evidence-based content includes the Listen-Empathize-Agree-Partner (LEAP) communication Program, and Acceptance and Commitment Therapy. The family psychoeducation classes are to take place at a designated AHS location.

Limitations and Conclusion:

The described protocol is one of the first attempts in the literature to evaluate an evidence-based intervention for carers of young adults with psychotic illness. The current study builds on others by incorporating psychoeducational elements, modules specific to the LEAP approach, and modules specific to ACT. Furthermore, the design of the study intends to gather longitudinal 24-month post-intervention data from carers and service users, including health service utilization data.

Several limitations must be considered with regards to this protocol. First, using a pre-post design the investigators cannot draw causal conclusions regarding the effect of the intervention. To address this limitation the investigators will use secondary data from health records as a non-equivalent control group for health utilization data. A second limitation is that participants self-select for the study, and may differ systematically from those who choose not to participate. For example, the sample will likely be biased towards families who are already supportive and involved in their young adults' care. The sample of young adults participating will be additionally biased because those who are especially unwell may be unable to participate. By comparing the health utilization data of the participants to the nonequivalent control group in a longitudinal design the investigators will gain some evidence to rule out history effects. Even with these limitations, the described design builds on existing knowledge of effective family psychoeducation groups and their long term effects on young adults experiencing psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Young adult service user is aged 17-27 at time of recruitment
* Young adult service user has had an admission or discharge from an Alberta Health Services or Covenant Health psychiatric unit for psychosis in the Edmonton Zone within previous 12-months

Exclusion Criteria:

* Not proficient in English
* Young adult service user has NOT had an admission or discharge from an Alberta Health Services or Covenant Health psychiatric unit for psychosis in the Edmonton Zone within previous 12-months

Ages: 17 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Family Burden Interview Schedule | Baseline-Day 0 (Pre-intervention)
  assesses overall burden of the family related to supporting a loved one with addiction and mental health concerns, including the following domains: financial, routines and activities, leisure, relationships, physical health, mental health
Family Burden Interview Schedule | 9-Week Follow-Up (Post-Intervention)
  assesses overall burden of the family related to supporting a loved one with addiction and mental health concerns, including the following domains: financial, routines and activities, leisure, relationships, physical health, mental health
Family Burden Interview Schedule | 6-Month Follow-Up (Post-Intervention)
  assesses overall burden of the family related to supporting a loved one with addiction and mental health concerns, including the following domains: financial, routines and activities, leisure, relationships, physical health, mental health
Family Burden Interview Schedule | 24-Month Follow-Up (Post-Intervention)
  assesses overall burden of the family related to supporting a loved one with addiction and mental health concerns, including the following domains: financial, routines and activities, leisure, relationships, physical health, mental health
Positive and Negative Symptom Schedule | Baseline-Day 0 (Pre-intervention)
  assesses overall symptom severity of service users, including 7 positive symptoms (e.g., hallucinations, grandiosity, etc.), 7 negative symptoms (e.g., blunted affect, emotional withdrawal) and general symptoms (e.g., anxiety, lack of judgement/insight, poor impulse control)
Positive and Negative Symptom Schedule | 9-Week Follow-Up (Post-Intervention)
  assesses overall symptom severity of service users, including 7 positive symptoms (e.g., hallucinations, grandiosity, etc.), 7 negative symptoms (e.g., blunted affect, emotional withdrawal) and general symptoms (e.g., anxiety, lack of judgement/insight, poor impulse control)
Positive and Negative Symptom Schedule | 6-Month Follow-Up (Post-Intervention)
  assesses overall symptom severity of service users, including 7 positive symptoms (e.g., hallucinations, grandiosity, etc.), 7 negative symptoms (e.g., blunted affect, emotional withdrawal) and general symptoms (e.g., anxiety, lack of judgement/insight, poor impulse control)
Positive and Negative Symptom Schedule | 24-Month Follow-Up (Post-Intervention)
  assesses overall symptom severity of service users, including 7 positive symptoms (e.g., hallucinations, grandiosity, etc.), 7 negative symptoms (e.g., blunted affect, emotional withdrawal) and general symptoms (e.g., anxiety, lack of judgement/insight, poor impulse control)
Manchester Short Assessment of Quality of Life | Baseline-Day 0 (Pre-intervention)
  assessing service user quality of life on a scale of 1 (couldn't be worse) to 7 (couldn't be better) and "yes/no" for select items.
Manchester Short Assessment of Quality of Life | 9-Week Follow-Up (Post-Intervention)
  assessing service user quality of life on a scale of 1 (couldn't be worse) to 7 (couldn't be better) and "yes/no" for select items.
Manchester Short Assessment of Quality of Life | 6-Month Follow-Up (Post-Intervention)
  assessing service user quality of life on a scale of 1 (couldn't be worse) to 7 (couldn't be better) and "yes/no" for select items.
Manchester Short Assessment of Quality of Life | 24-Month Follow-Up (Post-Intervention)
  assessing service user quality of life on a scale of 1 (couldn't be worse) to 7 (couldn't be better) and "yes/no" for select items.

SECONDARY OUTCOMES:
Inpatient Readmission Rate | 12-24 months post-intervention
  Readmission rate for mental health diagnosis within 30 days of an inpatient discharge
Inpatient Readmission Rate | 12-months pre-intervention
  Readmission rate for mental health diagnosis within 30 days of an inpatient discharge
Inpatient Readmission Rate | 12-months post-intervention
  Readmission rate for mental health diagnosis within 30 days of an inpatient discharge
Inpatient Admission Frequency | 12-months pre-intervention
  Frequency of hospital admissions for mental health diagnosis
Inpatient Admission Frequency | 12-months post-intervention
  Frequency of hospital admissions for mental health diagnosis
Inpatient Admission Frequency | 12-24 months post-intervention
  Frequency of hospital admissions for mental health diagnosis
Emergency Department Visit Frequency | 12-months pre-intervention
  Frequency of emergency departments visits within 30 days of last emergency presentation
Emergency Department Visit Frequency | 12-months post-intervention
  Frequency of emergency departments visits within 30 days of last emergency presentation
Emergency Department Visit Frequency | 12-24 months post-intervention
  Frequency of emergency departments visits within 30 days of last emergency presentation
Community Appointment Frequency | 12-months pre-intervention
  Appointment frequency for community-based services
Community Appointment Frequency | 12-months post-intervention
  Appointment frequency for community-based services
Community Appointment Frequency | 12-24 months post-intervention
  Appointment frequency for community-based services
Crisis Service Frequency | 12-months pre-intervention
  Frequency of crisis calls and visits
Crisis Service Frequency | 12-months post-intervention
  Frequency of crisis calls and visits
Crisis Service Frequency | 12-24 months post-intervention
  Frequency of crisis calls and visits

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Robles, md, Principal Investigator — University of Alberta; Adam Abba-Aji, MD, Principal Investigator — Alberta Health services
Locations (4):
- Canada (4):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Alberta Hospital Edmonton, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Yes
All IPD datasets that will be collected and analyzed for this study will be available by request from the corresponding author. Given the small study population, narrow geographic region of recruitment, and Alberta Health Services' data sharing policies, potentially identifying demographic data will not be available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available to requesting individuals/organizations through the corresponding author for a timeframe appropriate to the requesting party's needs.
Access Criteria: The purpose and timeframe of the requesting individuals/organizations dataset access will be reviewed on a case by case basis by the research team and is subject to approval by Alberta Health Services based on data sharing policies.

REFERENCES:
- [Background] Alberta Health Services. (2018). Patient and Family Centered Care Resource Kit: How to Improve the Patient Experience. Quality and Healthcare Improvement, Engagement and Patient Experience Department.
- [Background] Amador X. (2020).I Am Not Sick, I Don't Need Help! How To Help Someone Accept Treatment. New York: Vida Press
- [Background] American Psychological Association [APA]. (2011). Family Interventions. Retrieved on August 9, 2022 from https://www.apa.org/pi/about/publications/caregivers/practice-settings/intervention/family
- [Background] Day, K., & Petrakis, M. (2017). Family interventions in early psychosis service delivery: A systematized review. Social Work in Mental Health, 15(6): 632-650. doi:10.1080/15332985.2016.1271381
- [Background] Day K, Starbuck R, Petrakis M. Family group interventions in an early psychosis program: A re-evaluation of practice after 10 years of service delivery. Int J Soc Psychiatry. 2017 Aug;63(5):433-438. doi: 10.1177/0020764017710301. Epub 2017 May 24. PMID 28537124
- [Background] Early Psychosis Guidelines Writing Group and EPPIC National Support Program (2016). Australian Clinical Guidelines for Early Psychosis, 2nd edition update, Orygen, The National Centre of Excellence in Youth Mental Health, Melbourne.
- [Background] Ewertzon M, Hanson E. Support Interventions for Family Members of Adults with Mental Illness: A Narrative Literature Review. Issues Ment Health Nurs. 2019 Sep;40(9):768-780. doi: 10.1080/01612840.2019.1591547. Epub 2019 May 30. PMID 31145025
- [Background] Hayes, S.C., Strosahl, K.D., & Wilson, K.G. (1999)Acceptance and commitment therapy: An experiential approach to behavior change. Guilford Press.
- [Background] Jolley S, Johns LC, O'Donoghue E, Oliver J, Khondoker M, Byrne M, Butler L, De Rosa C, Leal D, McGovern J, Rasiukeviciute B, Sim F, Morris E. Group acceptance and commitment therapy for patients and caregivers in psychosis services: Feasibility of training and a preliminary randomized controlled evaluation. Br J Clin Psychol. 2020 Nov;59(4):524-551. doi: 10.1111/bjc.12265. Epub 2020 Sep 17. PMID 32944971
- [Background] Kreyenbuhl J, Buchanan RW, Dickerson FB, Dixon LB; Schizophrenia Patient Outcomes Research Team (PORT). The Schizophrenia Patient Outcomes Research Team (PORT): updated treatment recommendations 2009. Schizophr Bull. 2010 Jan;36(1):94-103. doi: 10.1093/schbul/sbp130. Epub 2009 Dec 2. PMID 19955388
- [Background] MacCourt, P. (2013). Family Caregivers Advisory Committee, Mental Health Commission of Canada. National Guidelines for a Comprehensive Service System to Support Family Caregivers of Adults with Mental Health Problems and Illnesses. Calgary, AB: Mental Health Commission of Canada. Retrieved from: http://www.mentalhealthcommission.ca
- [Background] McFarlane WR, Dixon L, Lukens E, Lucksted A. Family psychoeducation and schizophrenia: a review of the literature. J Marital Fam Ther. 2003 Apr;29(2):223-45. doi: 10.1111/j.1752-0606.2003.tb01202.x. PMID 12728780
- [Background] Poon, A.W.C., Curtis, J., Howard, A., Ward, P.B., & Lappin, J.M. (2019). Health of Carers of Young People with Early Psychosis: A Biopsychosocial Approach. Australian Social Work, 72(3): 260-273, DOI: 10.1080/0312407X.2018.1530269
- [Background] Rachamim L, Nacasch N, Sinay I. Complicated Grief, Depression, Health and Attachment Style in First Degree Relatives of Individuals with a Chronic Psychotic Disorders. Community Ment Health J. 2022 Apr;58(3):526-535. doi: 10.1007/s10597-021-00848-z. Epub 2021 Jun 16. PMID 34132930
- [Background] Rosas-Santiago, F.J., Genchi, J.J., Heredia, I.S., & Zamora, V.E.R. (2022). Psychoeducation and group acceptance and commitment therapy as psychological support strategies for informal caregivers of patients with a first psychotic episode: An experimental study. Psychosis: Psychological, Social and Integrative Approaches.[Preprint]. doi:10.1080/17522439.2022.2061041.
- [Background] World Health Organization. (2013). Mental health action plan 2013-2020. World Health Organization Library Cataloguing-in-Publication Data. https://www.who.int/publications/i/item/9789241506021
- [Derived] Zentner KE, Shettell K, Abba-Aji A, Robles M. Supporting patients by family education in psychotic illness: a longitudinal pre-post study protocol. BMJ Open. 2023 Oct 24;13(10):e072881. doi: 10.1136/bmjopen-2023-072881. PMID 37879701